CLINICAL TRIAL: NCT04377204
Title: The Utility of Long-acting Local Anesthetic Agents in Reducing Post-operative Opioid Requirements Following Rhinoplasty: A Multi-institutional, Randomized, Single Blinded Clinical Trial
Brief Title: The Utility of Long-acting Local Anesthetic Agents in Reducing Post-operative Opioid Requirements Following Rhinoplasty
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Our Lady of the Lake Hospital (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Leslie Son, Academic Research Director, Our Lady of the Lake Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OurLadyLH
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Pain, Postoperative; Local Anesthetic
Keywords: rhinoplasty; bupivacaine; pain management
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Intervention Model Description: Single blinded cohort intervention
Who Masked: Participant
Masking Description: Patients will be consented to participate, but will be blinded to which preoperative local anesthetic regimen they will receive for their rhinoplasty procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine Group (Active Comparator): Local injection of 1% lidocaine with 1:100,000 epinephrine one time pre-operatively prior to general anesthesia
  Interventions: Drug: Lidocaine
- Lidocaine with Bupivacaine (Active Comparator): Local injection of 1% lidocaine with 1:100,000 epinephrine mixed 1:1 with 0.5% marcaine bupivacaine with 1:200,000 epinephrine, one time pre-operatively prior to general anesthesia
  Interventions: Drug: marcaine bupivacaine

INTERVENTIONS:
Drug: marcaine bupivacaine — This drug is already FDA approved and used for the indication as a local anesthetic. The study herein would like to examine the pain outcomes of enrolled patients who will either have lidocaine alone OR lidocaine+bupivacaine combination locally prior to rhinoplasty surgery.
  Arms: Lidocaine with Bupivacaine
Drug: Lidocaine — This drug is already FDA approved and used for the indication as a local anesthetic. The study herein would like to examine the pain outcomes of enrolled patients who will either have lidocaine alone OR lidocaine+bupivacaine combination locally prior to rhinoplasty surgery.
  Arms: Lidocaine Group

SUMMARY:
On average, more than 130 Americans die every day from opioid overdose. Surgeons provide 37% of all opioid prescriptions in the United states, second only behind pain management physicians. A recent report found that patients who receive a 5-day supply of opioid medication have a 10% chance of using opioids 12 months later. Additionally, studies have shown that many opioid abusers are not the intended recipient, with over half diverting them from friends and family.

Rhinoplasty is one of the most common procedures performed by facial plastic surgeons, with over 215,000 performed in the United States in 2017. Patients undergoing nasal surgery have been shown to be at significant risk for persistent and prolonged opioid use after filling an opioid prescription in the perioperative period. Thus, the management of postoperative pain without contributing to the opioid epidemic is a imperative.

The first three days following nasal surgery are generally associated with considerable pain, with the highest levels occuring within the initial 24 hours. Published studies have demonstrated the benefit of non-opioid medications following rhinoplasty, such as pregabalin and celecoxib. There has also been growing recognition of the benefits of "pre-emptive analgesia," such as the use of local anesthesia, which not only helps control pain, but in turn decreases the anxiety caused by pain and can prevent patient turning to narcotics to break the cycle. These studies have predominantly focused on the immediate postoperative period, e.g. the first 24 hours.

Currently, many surgeons use lidocaine with 1% epinephrine as local anesthesia for rhinoplasty due to its widespread availability, rapid time to onset, and safety profile. Several studies have shown the benefit of Marcaine bupivacaine over lidocaine for pain control and opioid consumption during the first 24 hours after surgery. This is not surprising, as the half-life of lidocaine is approximately 90 minutes in a healthy individual, compared to 160 minutes for Marcaine bupivacaine. However, there are no studies to date that have evaluated the effect that long-acting local anesthesia has on post-operative opioid consumption past the first 24 hours after surgery. Our study aims to compare total postoperative opioid use for patients who received lidocaine as local anesthesia at the time of surgery versus a mixture of lidocaine and Marcaine bupivacaine.

DETAILED DESCRIPTION:
The local anesthesia regimen administered prior to surgery is a standard practice for rhinoplasty procedures. However, there is variation in the kind of anesthetic utilized during this time. In our practice, we have used different combinations along with epinephrine which include lidocaine or lidocaine with Marcaine bupivacaine dilutions. Although both are effective at pre-operative local numbing, investigators have seen less reported pain outcomes as perceived by the patient feedback. Therefore, investigators aim to identify specifically the usage of post-operative pain medication with those who had an epinephrine/lidocaine local anesthetic vs. those who had the epi/lidocaine/bupivacaine combination. Patients will be informed about the study and consented for participation. They will be randomized pre-operatively by permuted block assignment to the control treatment (1% lidocaine with 1:100,000 epinephrine) or the study treatment (1% lidocaine with 1:100,000 epinephrine mixed 1:1 with 0.5% Marcaine bupivacaine with 1:200,000 epinephrine) using a predetermined weight-calculated maximum dosage that would be safe for injection of either anesthesia.

As per standard procedure, the patients will be premedicated with a standardized dose of versed if determined necessary by anesthesia. Anesthesia will be induced utilizing weight based dosing of propofol and rocuronium. Intraoperative anesthesia will be maintained utilizing total intravenous anesthesia (propofol, fentanyl/remifentanyl doses). All patients will be given antibiotics (weight based dosing, Ancef or Clindamycin) and 8mg of dexamethasone prior to skin incision. Once anesthesia has been induced, the nose will be injected with local anesthesia as follows: transcutaneous to the bilateral dorsal nasal and the angular neurovascular bundles, transcutaneously along the columella and nasal dorsum, transnasally along the nasal dorsum and ala, the bilateral nasal septum, and the inferior turbinates with a total dose of 10ml's. Topical decongestion and anesthesia will then be obtained with 3 x 0.5cm cottonoids soaked with 4% cocaine placed bilaterally. A standard external rhinoplasty approach will the be performed, and grafting done as necessary. At then end of the procedure, Doyle nasal septal splints will be placed (Reuter-Bivalves if alar grafting performed).

In the immediate post-operative period, pain will be controlled with short acting analgesics (standardized regimen for all patients to be decided with anesthesia team) while in the acute care setting and recorded again as per standard of care. Once discharged from acute care, the patient will be given instructions to control their pain with acetaminophen (1000mg every 8 hours) scheduled during the first 72 hours, then as needed thereafter. They will also be given a prescription for oxycodone (15 tablets) with instruction to take 5mg every 6 hours as needed for breakthrough pain. They will be provided a pain diary for the first 24 hours to record their pain using the Faces scale (ranging 1-10 with 1 being no pain up to 10 being the worst pain ever experienced) at the 1, 2, 4, 6, 12, and 24 hours marks after discharge from surgery. Additionally, they will be asked to keep track of how many pain medications (oxycodone) they took over the first week after surgery. Their pain scores and amount of medication utilized will be recorded upon their follow up visit to the clinic.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 and over
* undergoing external rhinoplasty

Exclusion Criteria:

* Pre-existing chronic pain within 30 days prior to surgery
* Opioid use within 30 days before their surgery
* Patients undergoing a concurrent procedure (i.e. facial rejuvenation)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number and frequency of Pain pills taken up to 1 week post-op | 7 days post-operatively
  Patients will record the frequency and number of oxycodone pills taken for pain up to 7 days post-op

SECONDARY OUTCOMES:
Pain scores up to 24 hrs post-operatively | 24 hours
  Patients will be asked to maintain a pain diary to record their pain on a FACES scale at 1, 2, 4, 6, 12 and 24hrs post-operatively. The pain scale will be from 1-10 with 1 indicating no pain present up to a maximum score of 10 indicating the worst pain they've ever felt.

CONTACTS AND LOCATIONS:
Overall Officials: Justin C Sowder, MD, Principal Investigator — Louisiana State University Health Sciences Center - New Orleans
Locations (1):
- Our Lady of the Lake Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No